CLINICAL TRIAL: NCT05229549
Title: Open-label, Randomized, 4-way Crossover, Monocentric, Controlled Study to Evaluate the Effect on Nitrogen Retention of Two Different Posology Schemes of PKU GOLIKE PLUS 3-16 and Free AAs in Patients With Phenylketonuria
Brief Title: Study to Evaluate the Effect on Nitrogen Retention of Two Different Posology Schemes of PKU GOLIKE PLUS 3-16 and Free AAs in Patients With Phenylketonuria
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrolment
Sponsor: APR Applied Pharma Research s.a. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLK-2021
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2022-01

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A. One day treatment with 3 self-administrations of GOLIKE PLUS 3-16 (Active Comparator)
  Interventions: Other: GOLIKE PLUS 3-16
- B. One day treatment with 2 self-administrations of GOLIKE PLUS 3-16 (Active Comparator)
  Interventions: Other: GOLIKE PLUS 3-16
- C. One day treatment with 3 self-administrations of free AAs (Placebo Comparator)
  Interventions: Other: Free AAs
- D. One day treatment with 2 self-administrations of free AAs (Placebo Comparator)
  Interventions: Other: Free AAs

INTERVENTIONS:
Other: GOLIKE PLUS 3-16 — PKU GOLIKE PLUS 3-16 is a food for special medicinal purposes (FSMP) for the dietary management of PKU.
  Arms: A. One day treatment with 3 self-administrations of GOLIKE PLUS 3-16; B. One day treatment with 2 self-administrations of GOLIKE PLUS 3-16
Other: Free AAs — It is an immediate-release free AAs mixture with the same qualitative and quantitative composition of PKU GOLIKE PLUS 3-16.
  Arms: C. One day treatment with 3 self-administrations of free AAs; D. One day treatment with 2 self-administrations of free AAs

SUMMARY:
This is an open-label, randomized, 4-way crossover, monocentric, controlled study in patients (3 ≤ years of age ≤ 20 )) with phenylketonuria (PKU).

The primary comparison will be between the test product (PKU GOLIKE PLUS 3-16, a prolonged-release amino-acids (AAs) mixture) and the reference product (an immediate-release free AAs mixture with the same qualitative and quantitative composition of PKU GOLIKE PLUS 3-16). PKU GOLIKE PLUS 3-16 is a food for special medicinal purposes (FSMP) for the dietary management of PKU.

The study will consist of a screening visit (T0), four test days taking place on Sunday (T1-T4), each separated by a washout period (a period of time when a participant is taken off a treatment in order to eliminate its effects) and with the study products being self-administered at home, and a final visit (T5).

Following informed consent and verification of eligibility criteria, 24 patients with PKU will be randomized in a 1:1:1:1 ratio to one of the four randomization sequences ABCD, BDAC, DCBA or CADB.

A, B, C and D will be:

A. One day treatment with 3 self-administrations of GOLIKE PLUS 3-16 (1.2 g/kg total daily dose of AA) B. One day treatment with 2 self-administrations of GOLIKE PLUS 3-16 (1.2 g/kg total daily dose of AA) C. One day treatment with 3 self-administrations of free AAs (1.2 g/kg total daily dose of AA) D. One day treatment with 2 self-administrations of free AAs (1.2 g/kg total daily dose of AA)

GOLIKE PLUS 3-16 and the free AAs mixture will be the only protein substitute allowed on each test day, and no sports activities will be allowed on the test days.

24-hour urines and five blood spots will be collected on each test day. A patient's diary will be used to collect information on patient compliance, 24-hour urines and blood spot collections, diet, daily activities, adverse events and concomitant medications.

Patients completing all four test days will be asked to go to the center for a final visit (T5) taking place within 2 weeks from the last product administration.

DETAILED DESCRIPTION:
This is an open-label, randomized, 4-way crossover, monocentric, controlled study in patients (3 ≤ years of age ≤ 20 ) with phenylketonuria (PKU).

The primary comparison will be between the test product (PKU GOLIKE PLUS 3-16, a prolonged-release amino-acids (AAs) mixture, in this protocol referred to as GOLIKE PLUS 3-16) and the reference product (an immediate-release free AAs mixture with the same qualitative and quantitative composition of PKU GOLIKE PLUS 3-16). PKU GOLIKE PLUS 3-16 is a food for special medicinal purposes (FSMP) for the dietary management of PKU.

The study will consist of a screening visit (T0), four test days taking place on Sunday (T1-T4), each separated by a washout period (a period of time when a participant is taken off a treatment in order to eliminate its effects) and with the study products being self-administered at home, and a final visit (T5). A telephone call will be made to the patients during each washout period. Test days will occur preferably on four consecutive weeks with a 1-week washout period between each test day. Washout can be extended up to 2 weeks in case a dose delay (i.e. delay of the test day) is deemed necessary.

Following informed consent and verification of eligibility criteria, 24 patients with PKU will be randomized in a 1:1:1:1 ratio to one of the following four randomization sequences: ABCD, BDAC, DCBA or CADB.

A, B, C and D will be:

A. One day treatment with 3 self-administrations of GOLIKE PLUS 3-16 (1.2 g/kg total daily dose of AA) B. One day treatment with 2 self-administrations of GOLIKE PLUS 3-16 (1.2 g/kg total daily dose of AA) C. One day treatment with 3 self-administrations of free AAs (1.2 g/kg total daily dose of AA) D. One day treatment with 2 self-administrations of free AAs (1.2 g/kg total daily dose of AA) No change in the randomization sequence will be allowed. Diet will be standardized among different patients in terms of calories and nutrients ranges on each test day, according to the age and body weight of the patients. Moreover, the type of food ingested in 24 hours will be the same on each test day in the same patient.

GOLIKE PLUS 3-16 and the free AAs mixture will be the only protein substitute allowed on each test day, and no sports activities will be allowed on the test days.

24-hour urines and five blood spots will be collected on each test day. Timing of self-administrations, meals and blood spots will be defined for each test day. On the test days, no food will be allowed outside of the defined time windows. The first self-administration of each test day will be performed after overnight fasting (10 -12 h) and before any food intake takes place. Urine should be voided before the first self-administration and not collected. 24-hour urine collection begins thereafter.

The day after each test day a designated courier will collect urine samples and blood spots at the patient's home and will bring them to the center.

A patient's diary will be used to collect information on patient compliance, 24-hour urines and blood spot collections, diet, daily activities, adverse events and concomitant medications.

Adverse events will be continuously monitored during the study, starting from informed consent. Adverse events will be collected by the patients (or by a parent/guardian) in the diary and during the telephone calls made by the Investigator to the patients. Moreover, patients (or parents/guardians) will be instructed to promptly report adverse events occurring during the study to the Investigator.

Patients completing all four test days will be asked to go to the center for a final visit (T5) taking place within 2 weeks from the last product administration. Patients prematurely discontinued from the study will be asked to attend a discontinuation visit possibly taking place within 2 weeks from the last product administration. At the final/discontinuation visit, patients will be asked to return their diaries and the Investigator will verify all information reported in the patient's diary and record it in the electronic Case Report Form (eCRF).

ELIGIBILITY:
Inclusion Criteria:

1. Signed, informed consent obtained prior to being enrolled into the study and prior to starting any data collection. Consent of a legally authorized guardian is required for legally minor patients as defined by local regulation. If the patient is legally a minor, signed written consent shall be obtained from parent(s)/legal guardian and assent obtained from the patient, if applicable.
2. Male or female, aged 3-20 (limits included).
3. Patients with diagnosis of PKU at newborn screening.
4. Patients starting low Phe diet before 1 month of age.
5. Ability and willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

1. Known or suspected hypersensitivity to any excipients/components of the investigational products.
2. Treatment with therapy for PKU other than amino-acids supplementation.
3. Patients aged >12 years old with 4 repeated average values of blood Phe >600 µM in the previous 6 months.
4. Patients aged <12 years old with 4 repeated average values of blood Phe >360 µM in the previous 6 months.
5. Any moderate to severe medical condition, which in the opinion of the Investigator would interfere with the study procedures or study outcome (reasoning to be provided), such as history of clinically significant diseases or malfunctions including, but not limited to, gastrointestinal, renal, hepatic, pulmonary, cardiovascular or endocrine disease, hemophilia, hyperlipidemia, impaired glucose tolerance or diabetes (type 1 or 2), or anemia.
6. History of poor co-operation, non-compliance with medical treatments and diet, or poor adherence to investigational procedures.
7. Any current participation in another clinical trial involving investigational or marketed products in the 3 months prior to the inclusion in this study.
8. Pregnancy or lactation.

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Difference of GOLIKE PLUS 3-16 versus free AAs in terms of nitrogen retention after one day of product intake | Over 24 hours of each test day.
  Nitrogen excretion in the 24-hour urines of each test day is measured.

SECONDARY OUTCOMES:
Comparison of impact of 2 self-administrations of GOLIKE PLUS 3-16 and of 3-self administrations of free AAs on nitrogen retention after one day of product intake | Over 24 hours of each test day.
  Nitrogen excretion in the 24-hour urines of each test day is measured.
Comparison of the impact of 2 self-administrations of GOLIKE PLUS 3-16 and of 3 self-administrations of GOLIKE PLUS 3-16 on nitrogen excretion | Over 24 hours of each test day.
  Nitrogen excretion in the 24-hour urines of each test day is measured.
Comparison of the the impact of GOLIKE PLUS 3-16 and of free AAs on phenylalanine (Phe) and tyrosine (Tyr) levels in blood on each test day. | Over 24 hours of each test day.
  Levels of Phe and Tyr in blood at pre-defined time points

OTHER OUTCOMES:
Comparison of the impact of GOLIKE PLUS 3-16 and of free AAs on branched-chained amino acids (leucine, isoleucine, valine) levels in blood on each test day. | Over 24 hours of each test day.
  Levels of branched-chained amino acids (leucine, isoleucine, valine) in blood at pre-defined time points
Comparison of the impact of GOLIKE PLUS 3-16 and of free AAs on the urinary creatinine/height index after one day of product intake. | Over 24 hours of each test day.
  Urinary creatinine/height index in the 24-hour urines of each test day.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Banderali, Principal Investigator — ASST Santi Paolo e Carlo, Presidio Ospedale San Paolo, Via Antonio di Rudinì 8 - 20142, Milano (Italy)
Locations (1):
- San Paolo Hospital, Milan, Italy